CLINICAL TRIAL: NCT01560377
Title: Open Label Clinical Study to Demonstrate the Utility of Intra-operative Perfusion Assessment Using NIR Fluorescence Angiography With the PINPOINT® Endoscopic Fluorescence Imaging System and to Assess the Impact of PINPOINT on the Surgical Decision Making Process and on Surgical Outcomes in Laparoscopic Left Anterior Resection Procedures
Brief Title: Perfusion Assessment in Laparoscopic Left Anterior Resection
Acronym: PILLAR II
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novadaq Technologies ULC, now a part of Stryker (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Version 1
Record Dates: First submitted 2012-03-19; First posted 2012-03-22 (Estimated); Results first posted 2018-10-29 (Actual); Last update posted 2018-12-11 (Actual); Status verified 2018-11

CONDITIONS: Rectal Cancer; Colon Cancer; Crohn's Disease; Polyp; Procidentia; Diverticulitis
Keywords: Laparoscopic low anterior colon resection; Laparoscopic left colectomy; Colectomy; Rectal cancer; Colon cancer; Crohn's Disease; Polyp; Procidentia; Diverticulitis
MeSH Terms: conditions — Rectal Neoplasms; Colonic Neoplasms; Crohn Disease; Polyps; Prolapse; Diverticulitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Subjects Imaged with PINPOINT (Experimental): Colonic tissue perfusion assessed with PINPOINT for laparoscopic left colectomy in the lower tract.
  Interventions: Device: PINPOINT Endoscopic Fluorescence Imaging System

INTERVENTIONS:
Device: PINPOINT Endoscopic Fluorescence Imaging System — The PINPOINT system will be used to provide real-time endoscopic visible and endoscopic NIR fluorescence imaging. PINPOINT enables surgeons to perform routine visible light endoscopic procedures as well as further visually assess vessels, blood flow and related tissue perfusion with near infra-red imaging during minimally invasive surgery

SUMMARY:
The purpose of this study is to demonstrate that NIR fluorescence angiography using the PINPOINT Endoscopic Fluorescence Imaging System ("PINPOINT System" or "PINPOINT") can assess viability of colon tissue during laparoscopic left colectomy. This information will provide the surgeon with clinically relevant information in assessing whether or not the tissue has adequate blood supply in the lower section of the colon prior to a colectomy.

DETAILED DESCRIPTION:
Colectomy is a surgical procedure in which a part or all of the colon is removed. It is used to treat a variety of diseases including colon cancer, diverticulitis, inflammatory bowel disease (including ulcerative colitis or Crohn's disease) and infarcted bowel.

This study is the second phase of a three phase process to demonstrate the clinical utility of perfusion assessment by NIR fluorescence angiography in colectomy. The initial phase (Phase I) consisted of a number of small investigative studies that have now been completed. Upon successful completion of this study, it is anticipated that a prospective, multi center, randomized trial will be conducted (Phase III). Information learned from this present study will help guide the design of the randomized trial e.g. specific patient populations that may best benefit from this imaging modality and how randomization should be conducted (e.g. imaged cohort vs. non imaged, or all subjects imaged but then randomized to no image assessment in one arm of the study).

ELIGIBILITY:
Inclusion Criteria:

* Subject is scheduled for laparoscopic left colectomy in the lower region (planned anastomosis located 5 - 15 cm from anal verge)
* A negative pregnancy test for women of childbearing potential prior to surgery

Exclusion Criteria:

* Subject has a previous history of adverse reaction or known allergy to ICG, iodine or iodine dyes
* Subject has any medical condition, which in the judgment of the Investigator and/or designee makes the subject a poor candidate for the investigational procedure
* Subject is a pregnant or lactating female

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2012-05; Primary Completion 2013-10 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Stamos, MD, Principal Investigator — University of California, Irvine
Locations (11):
- United States (11):
  - University of Southern California, Los Angeles, California
  - University of California, Irvine, Orange, California
  - University of California San Diego, San Diego, California
  - University of California San Francisco, San Francisco, California
  - Cleveland Clinic Florida, Weston, Florida
  - Ochsner Medical Center, New Orleans, Louisiana
  - Mayo Clinic, Rochester, Minnesota
  - Maimonides Medical Center, Brooklyn, New York
  - Beth Israel Medical Center, New York, New York
  - Weill Cornell Medical College, New York, New York
  - University Hospital Case Medical Center, Cleveland, Ohio

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 147 patients were enrolled, of whom 139 were eligible for analysis. Patients were enrolled at 11 centers in the United States.
Period: Overall Study
Arm/Group | Subjects Imaged With PINPOINT
Started | 147
Eligible for Analysis | 139
Completed | 147
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Patients undergoing left colectomy/low anterior resection
Arm/Group | Subjects Imaged With PINPOINT
Number analyzed (Participants) | 139
Age, Continuous [Mean (Full Range); unit: years] | 58 [44 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65
  Male | 74
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10
  Not Hispanic or Latino | 129
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 14
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 106
  More than one race | 0
  Unknown or Not Reported | 12
Region of Enrollment [Number; unit: participants]
  United States | 139
ASA Classification (American Society of Anesthesiologists) [Count of Participants; unit: Participants]
  I (normal healthy patient) | 17
  II (patient with mild systemic disease) | 73
  III (patient with severe systemic disease) | 46
  IV (severe life threating systemic disease) | 3
BMI [Count of Participants; unit: Participants]
  BMI > 30 kg/m^2 | 42
  BMI < 30 kg/m^2 | 97
Preoperative chemotherapy [Count of Participants; unit: Participants]
  Yes | 13
  No | 126
Preoperative radiation therapy [Count of Participants; unit: Participants]
  Yes | 15
  No | 124
Diagnosis [Count of Participants; unit: Participants]
  Diverticulitis | 61
  Rectal cancer | 35
  Colon cancer | 29
  Polyp | 6
  Procidentia | 4
  Crohn's disease | 1
  Colovesical fistula | 1
  Radiation stricture | 1
  Sigmoid volvulus | 1

OUTCOME MEASURES:

1. Primary Outcome: PINPOINT System Utility in Left Colectomy Surgery
Description: To demonstrate the utility of intra-operative assessment of colon perfusion, using the PINPOINT System to optimize the location at which to transect the colon in laparoscopic left colectomies and to assess mucosal perfusion of the completed anastomosis following proximal anastomosis in laparoscopic left colectomy.
Time Frame: Day of Operation - Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Subjects Imaged With PINPOINT
Number analyzed (Participants) | 139
Participants
  Change to surgical plan due to Fluorescence | 11
  No change to surgical plan due to Fluorescence | 128

2. Secondary Outcome: Safety of the PINPOINT System
Description: To assess safety related outcomes of the laparoscopic left colectomies with intra-operative assessment of perfusion using the PINPOINT Endoscopic Fluorescence Imaging System for guidance.
Time Frame: Through hospital discharge or at 30 days post procedure, whichever is later
Measure: Count of Participants; unit: Participants
Arm/Group | Subjects Imaged With PINPOINT
Number analyzed (Participants) | 139
Participants
  Clinical anastomotic leak & confirmed by radiology | 2
  Post-operative fever | 7
  Delay in return of bowel function | 5
  No major post-operative clinical complication | 125

ADVERSE EVENTS:
Arm/Group | Subjects Imaged With PINPOINT
Serious Adverse Events (participants affected / at risk) | 23/139
Other Adverse Events (participants affected / at risk) | 0/139
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Subjects Imaged With PINPOINT (N=139)
Anastomotic leak (Surgical and medical procedures) | 2
Pelvic abscess (Infections and infestations) | 2
Abdominal wall infection (Infections and infestations) | 1
Acute renal failure (Renal and urinary disorders) | 1
Blood transfusion (Blood and lymphatic system disorders) | 1
C. difficile colitis (Infections and infestations) | 2
Fever (General disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Ileus requiring nasogastric tube (Gastrointestinal disorders) | 1
Small bowel obstruction (Gastrointestinal disorders) | 1
Incisional hernia (Gastrointestinal disorders) | 1
Thrombosed left renal artery (Vascular disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Urinary tract infection (Renal and urinary disorders) | 1
Wound infection (Infections and infestations) | 1
Hypertension (Cardiac disorders) | 1
Hypokalemia (Hepatobiliary disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less